CLINICAL TRIAL: NCT05892133
Title: Prehabilitation Effect on Function and Patient Satisfaction Following Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 522685
Record Dates: First submitted 2023-05-03; First posted 2023-06-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-06

CONDITIONS: Prehabilitation; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal strength training (Experimental): eight weeks of leg press strength training prior to knee surgery
  Interventions: Behavioral: Maximal strength training
- Control (No Intervention): treatment as usual prior to knee surgery

INTERVENTIONS:
Behavioral: Maximal strength training — 3 sessions/ week. leg press at ~85% of one repetition maximum for 8 weeks
  Arms: Maximal strength training

SUMMARY:
Knee arthrosis has a high prevalence. Non-surgical treatment, such as exercise, is the first choice of treatment. However, most patients end up having a surgical procedure such as total knee arthroplasty. Following surgery with total knee replacement as much as 20% of patients report to not be satisfied with the results. It is noteworthy that this level of dissatisfaction has persisted over the last decades despite formidable progress in surgical methods and technology. Leg strength prior to surgery is associated with faster recovery post operatively, which may influence satisfaction. The investigators aim is to implement a period of strength training prior to surgery to evaluate if training prior to surgery may reduce the level of dissatisfaction post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Knee artrosis, refered to surgery

Exclusion Criteria:

* Kognitive disability
* Inflamatory disease in muscles
* varus/ valgus and extension deficit >15 degrees
* Neurological disorders

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Leg press strength | Baseline, 1 week pre-surgery, 3week post-surgery, 12 months post-surgery.
  The maximal weight that can be lifted once
Group differences in Patient satisfaction | Change from 3 week post-surgery, 12 months post-surgery.
  Satisfied with the results of knee surgery: yes/no

SECONDARY OUTCOMES:
Change in Voluntary activation | Baseline, 1 week pre-surgery, 3week post-surgery.
  Force production of thigh muscle during contraction with superimposed electrical stimulation
Change in Self reported knee function | Baseline, 1 week pre-surgery, 3week post-surgery, 12 months post-surgery.
  The Knee Injury and Osteoarthritis Outcome Score - Physical Function - Short Form
Change in Walking speed | Baseline, 1 week pre-surgery, 3week post-surgery, 12 months post-surgery.
  10 meter walking test
Change in Chair rising ability | Baseline, 1 week pre-surgery, 3week post-surgery, 12 months post-surgery.
  30 second sit to stand test
Change in Balance | Baseline, 1 week pre-surgery, 3week post-surgery, 12 months post-surgery.
  unipedal stance test, postural sway

CONTACTS AND LOCATIONS:
Overall Officials: Berg, Principal Investigator — Molde UC
Locations (1):
- Molde University College, Molde, Møre og Romsdal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izadi M, Toien T, Ohrn FD, Schnell Husby O, Kvitland Schnell Husby V, Bjorgen Winther S, Sherman R, Forsberg Brobakken M, Wang E, Berg OK. Effects of preoperative maximal strength training on muscle strength and function in total knee arthroplasty: A randomized controlled trial. Ann Phys Rehabil Med. 2026 Jan 13;69(2):102067. doi: 10.1016/j.rehab.2025.102067. Online ahead of print. PMID 41534474